CLINICAL TRIAL: NCT01298336
Title: Efficacy of Clarithromycin or Moxifloxacin Containing Regimen in 6 Months Sputum Conversion of Mycobacterium Xenopi
Brief Title: Treatment of Mycobacterium Xenopi Pulmonary Infection
Acronym: CAMOMY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PHRCN10-DR-ANDREJAK-MELLE
Record Dates: First submitted 2011-02-15; First posted 2011-02-17 (Estimated); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Atypical; Mycobacterium, Pulmonary, Tuberculous
Keywords: Mycobacterium Xenopi Pulmonary Infection; Clarithromycin; Moxifloxacin
MeSH Terms: conditions — Mycobacterium Infections; Latent Tuberculosis | interventions — Clarithromycin; Moxifloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Clarithromycin (Experimental)
  Interventions: Drug: Clarithromycin
- Moxifloxacin (Experimental)
  Interventions: Drug: Moxifloxacin

INTERVENTIONS:
Drug: Clarithromycin — 500 mg twice a day seven days a week
  Other Names: ZECLAR, NAXY
  Arms: Clarithromycin
Drug: Moxifloxacin — 400 mg per day seven days a week
  Other Names: IZILOX
  Arms: Moxifloxacin

SUMMARY:
The purpose of this study is to determine the 6-months sputum conversion rate with a clarithromycin or moxifloxacin containing regimen in patients with a M. xenopi pulmonary infection.

DETAILED DESCRIPTION:
In France, Mycobacterium xenopi is the second non-tuberculous mycobacteria responsible of pulmonary infections. There are few data in the literature regarding its treatment apart from two small randomized trials (42 and 34 patients, respectively) and a French retrospective study (136 patients). So, we decided to conduct a prospective randomized multicenter study to evaluate two treatment regimens for Mycobacterium xenopi pulmonary infection in 6-months sputum conversion.

Main objective: To determine the 6-months sputum conversion rate with a clarithromycin or moxifloxacin containing regimen in patients with M.xenopi pulmonary infections according to ATS / IDSA 2007 criteria.

Secondary Objectives: To compare the rate of sputum conversion after 3 and 6 months of treatment the clinical and radiological outcome and the 12 months mortality.

primary endpoint : Result of culture of respiratory samples 6 months after starting treatment.Culture samples taken 6 months after starting treatment against M. xenopi is either positive (presence of M. xenopi colonies with or without smear positive) or negative with smear and culture negative (see data collection and measurement methods).

Study plan: Any patient with at least one positive pulmonary M. xenopi sample may be eligible. If the patient underwent ATS / IDSA 2007 criteria of M. xenopi pulmonary infection (after clinical , radiological and microbiological evaluation), in the absence of exclusion criteria, the patient will be randomized to one of the two treatment arms (rifampicin+ ethambutol + clarithromycin or rifampicin + ethambutol + moxifloxacin). A clinical, radiological, microbiological and pharmacological monitoring will be done for each randomized patient. The recommended treatment duration is 12 months after conversion with a maximum duration of 18 months.

Number of patients required: This is a prospective randomized study with 2 parallel groups. The primary endpoint is considered for the whole study population. For an α risk of 5%, an accuracy of 10%, an expected conversion rate of 70% a total of 80 patients is required . For a 15% rate of non evaluable patients (died, lost of follow-up) we need to include 92 patients.

Study Duration: Inclusion for 24 months with a minimum follow-up of 6 months (to meet the main objective), and if possible a follow-up of 12 months per patient to meet the overall objectives of the study.

Prospects: To establish new treatment recommendations for M.xenopi pulmonary infection, based on microbiological and clinical efficacy criteria and tolerance criteria.

ELIGIBILITY:
Inclusion Criteria:

* The patient and/or legal representative of the patient has provided a written informed consent before inclusion in the study
* The patient is aged 18 or older
* The patient has signs of functional respiratory (cough, sputum, hemoptysis, dyspnea, chest pain and / or general signs (asthenia and / or anorexia and / or weight loss)
* The patient has a creatinine clearance above 30 ml / min
* The patient underwent a thoracic scan not older than one month before the first positive bacteriological sample.
* The patient underwent a bronchoscopy with sampling conducted in the territory corresponding to the radiographic
* The most plausible alternative diagnostics have been eliminated using the thoracic scan and bronchoscopy
* The patient has at least two positive cultures for M. xenopi sputum collected on two separate days AND/OR a positive culture for M. xenopi in a bronchoalveolar lavage or bronchial aspiration directed AND / OR transbronchial biopsy or lung biopsy with surgical histology for a mycobacterial infection (granuloma or Ziehl positive) and a culture positive M. xenopi, AND / OR biopsy with histology compatible with mycobacteriosis and one or more positive sputum culture for M . xenopi
* The patient is willing and able to take the study treatment throughout the duration
* If this is a woman of childbearing age, the patient is ready to use for the duration of the test contraception method other than estrogen-progestin
* The patient did not participate in another study evaluating an investigational drug within 30 days prior to enrollment in the study and agrees not to participate in another study for the duration of the study
* The patient is informed by the doctor and agreed that its data are processed in this study
* The patient understands / reads French and has no difficulty understanding the objectives of the study
* The patient has health insurance coverage

Exclusion Criteria:

* Hypersensitivity to any of the molecules (rifampicin, ethambutol, moxifloxacin, clarithromycin)
* Any patient with a relapse of a lung infection with M. xenopi
* The patient is treated with molecules that can interfere with cytochrome P450 and can not be replaced by another therapeutic class
* The patient is treated by prolonging the QT molecules which can not be replaced by another therapeutic class
* The patient is treated with alkaloid of ergot, cisapride, biperidil, pimozide, mizolastine
* The patient has heart failure with left ventricular ejection fraction below 30%
* Discovered on the balance sheet or history, we find that the patient infection with human immunodeficiency virus HIV 1 and 2 a long QT on ECG and / or arrhythmias or clinically significant bradycardia judged by the investigator cytolysis with transaminases increase more than 5 times normal renal failure with creatinine clearance below 30 ml / min
* The patient has cirrhosis Child Pugh C and / or porphyria
* There pregnancy or during breastfeeding
* The patient has an inability to meet the protocol requirements, including active substance abuse, according to the investigator.
* The patient has a history of tendinopathy with a fluoroquinolone
* The patient has a congenital galactosemia, malabsorption of glucose and galactose, or lactase deficiency
* The patient has a NORB (abnormalities of the visual field or color vision tested by an eye examination prior)
* Any other situation that, in the opinion of the investigator, would imply that participation in the study is not in the interest of the patient
* There is a risk of difficulty of monitoring, such as imminent transfer to a different region or country

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2011-03-02 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Sputum conversion at 6 months under three antibiotics treatment (Rifampin, ethambutol and a third drug clarithromycin or moxifloxacin) | 6 months
  Results of the smear and culture of three respiratory samples after 6 months of treatment.

SECONDARY OUTCOMES:
Sputum conversion at 3, 6, 9 and 12 months of treatment in the two different arms (clarithromycin containing regimen versus moxifloxacin containing regimen | 12 months
  At each endpoint (3, 6, 9 and 12 months), respiratory sample will be analyzed (smear and culture) to answer the second objective (to compare microbiological efficacy of clarithromycin-containing regimen versus moxifloxacin-containing regimen)
Clinical and radiological outcome after 3, 6 and 12 months of treatment according to the treatment arm | 12 months
  At each end-point (3, 6 and 12 months) :
  * clinical evaluation with analogic scale (sputum, cough, dyspnea, chest pain, hemoptysis) and weight
  * radiological evaluation: comparison of the size and number of lesions at each endpoint with basal data
Mortality after 12 months of treatment in the two compared regimen | 12 months
  Mortality status will be evaluated after 12 months of treatment. In case of deaths under treatment, the date will be collected. Comparative survival analysis will be realized between the two arms of treatment
Gastrointestinal toxicity and hematotoxicity after 1- 3- 6- 9- 12- months of treatment | 12 months
  At each end point (1- 3- 6- 9- 12 months), Rhodes score (gastro-intestinal tolerance)and WHO score for hematological, and gastrointestinal toxicity will be collected in the two arms

CONTACTS AND LOCATIONS:
Overall Officials: Claire ANDREJAK, Dr, Study Director — Centre Hospitalier Universitaire, Amiens; Claire ANDREJAK, MD, Principal Investigator — CHU Amiens; Vincent JOUNIEAUX, MD PhD, Principal Investigator — CHU Amiens; Nicolas VEZIRIS, MD-PhD, Principal Investigator — APHP Pitie Salpetriere Hospital, National Center Of Mycobacteria; Jacques CADRANEL, MD PhD, Principal Investigator — Tenon Hospital APHP Paris; Francois-Xavier LESCURE, MD, Principal Investigator — Tenon hospital APHP Paris
Locations (52):
- France (52):
  - CH Compiègne, Compiègne, Compiègne
  - CH Intercommunal Meulan, Les Mureaux, Les Mureaux
  - Centre National de Reference Des Mycobactéries, Paris, PARIS
  - CH Saint-Nazaire, Saint-Nazaire, Saint-Nazaire
  - CH Troyes, Troyes, Troyes
  - CH Abbeville, Abbeville
  - CHU Amiens, Amiens
  - CHU Angers, Angers
  - CH Argenteuil, Argenteuil
  - CHU Besançon, Besançon
  - CH Béthune, Béthune
  - Assistance Publique Hôpitaux de Paris CHU Avicenne, Bobigny
  - CHU Brest La Cavale, Brest
  - CHU Caen, Caen
  - CH Cannes, Cannes
  - CHU Clermont Ferrand Hôpital Gabriel Mont pied, Clermont-Ferrand
  - CH Sud Francilien, Corbeil-Essonnes
  - Centre Intercommunal de Créteil, Créteil
  - CHU Dijon, Dijon
  - CH Gonesse, Gonesse
  - CHU Grenoble, Grenoble
  - Assistance Publique Hôpitaux de Paris Hôpital Bicetre, Le Kremlin-Bicêtre
  - CH Le MANS, Le Mans
  - CHU Lille Hôpital Calmette, Lille
  - CHU Limoges Hôpital de Cluzeau, Limoges
  - CHU Lyon Hôpital La Croix Rousse, Lyon
  - Hopital Saint-Joseph, Marseille
  - Assistance Publique Hôpitaux de Marseille, Marseille
  - CHU Montpellier Hôpital Arnaud de Villeneuve, Montpellier
  - CHU Nantes, Nantes
  - CHU Nice, Nice
  - Chr Orleans, Orléans
  - Assistance Publique Hôpitaux de Paris Hôpital Saint Louis, Paris
  - Assistance Publique Hôpitaux de Paris Hôpital Saint Antoine, Paris
  - Assistance Publique Hôpitaux de Paris Hôpital BICHAT, Paris
  - Assistance Publique Hôpitaux de Paris, hôpital TENON, Paris
  - CHU Bordeaux Hôpital Haut Leveque, Pessac
  - CHU Poitiers, Poitiers
  - Hopital René DUBOS, Pontoise
  - CHU Reims, Reims
  - CHU de Rennes Hôpital Ponchaillou, Rennes
  - CH de Roubaix, Roubaix
  - CHU Rouen, Rouen
  - CHU de Saint Etienne, Saint-Etienne
  - CH de Saint Quentin, Saint-Quentin
  - CHU de Strasbourg, Strasbourg
  - Hôpital FOCH, Suresnes
  - CHU Toulouse, Toulouse
  - CH de Tourcoing, Tourcoing
  - CHU Tours Hôpital BRETONNEAU, Tours
  - CH de Valenciennes, Valenciennes
  - CHU Nancy, Vandœuvre-lès-Nancy

REFERENCES:
- [Background] Song JH, Yoon SY, Park TY, Heo EY, Kim DK, Chung HS, Lee JK. The clinical impact of drug-induced hepatotoxicity on anti-tuberculosis therapy: a case control study. Respir Res. 2019 Dec 16;20(1):283. doi: 10.1186/s12931-019-1256-y. PMID 31842883
- [Background] TIMPE A, RUNYON EH. The relationship of atypical acid-fast bacteria to human disease; a preliminary report. J Lab Clin Med. 1954 Aug;44(2):202-9. No abstract available. PMID 13184228
- [Background] RUNYON EH. Anonymous mycobacteria in pulmonary disease. Med Clin North Am. 1959 Jan;43(1):273-90. doi: 10.1016/s0025-7125(16)34193-1. No abstract available. PMID 13612432
- [Background] Griffith DE, Aksamit T, Brown-Elliott BA, Catanzaro A, Daley C, Gordin F, Holland SM, Horsburgh R, Huitt G, Iademarco MF, Iseman M, Olivier K, Ruoss S, von Reyn CF, Wallace RJ Jr, Winthrop K; ATS Mycobacterial Diseases Subcommittee; American Thoracic Society; Infectious Disease Society of America. An official ATS/IDSA statement: diagnosis, treatment, and prevention of nontuberculous mycobacterial diseases. Am J Respir Crit Care Med. 2007 Feb 15;175(4):367-416. doi: 10.1164/rccm.200604-571ST. No abstract available. PMID 17277290
- [Background] Falkinham JO 3rd. Nontuberculous mycobacteria in the environment. Clin Chest Med. 2002 Sep;23(3):529-51. doi: 10.1016/s0272-5231(02)00014-x. PMID 12370991
- [Background] von Reyn CF, Waddell RD, Eaton T, Arbeit RD, Maslow JN, Barber TW, Brindle RJ, Gilks CF, Lumio J, Lahdevirta J, et al. Isolation of Mycobacterium avium complex from water in the United States, Finland, Zaire, and Kenya. J Clin Microbiol. 1993 Dec;31(12):3227-30. doi: 10.1128/jcm.31.12.3227-3230.1993. PMID 8308115
- [Background] Smith MJ, Citron KM. Clinical review of pulmonary disease caused by Mycobacterium xenopi. Thorax. 1983 May;38(5):373-7. doi: 10.1136/thx.38.5.373. PMID 6879487
- [Background] Banks J, Hunter AM, Campbell IA, Jenkins PA, Smith AP. Pulmonary infection with mycobacterium xenopi: review of treatment and response. Thorax. 1984 May;39(5):376-82. doi: 10.1136/thx.39.5.376. PMID 6740540
- [Background] American Thoracic Society. Diagnosis standards and classification of tuberculosis and other mycobacterial diseases. New York: American Lung Association, 1974:25
- [Background] Diagnosis and treatment of disease caused by nontuberculous mycobacteria. Am Rev Respir Dis. 1990 Oct;142(4):940-53. doi: 10.1164/ajrccm/142.4.940. No abstract available. PMID 2282111
- [Background] Diagnosis and treatment of disease caused by nontuberculous mycobacteria. This official statement of the American Thoracic Society was approved by the Board of Directors, March 1997. Medical Section of the American Lung Association. Am J Respir Crit Care Med. 1997 Aug;156(2 Pt 2):S1-25. doi: 10.1164/ajrccm.156.2.atsstatement. PMID 9279284
- [Background] Subcommittee OT. Management of opportunist mycobacterial infections: Joint Tuberculosis Committee Guidelines 1999. Subcommittee of the Joint Tuberculosis Committee of the British Thoracic Society. Thorax. 2000 Mar;55(3):210-8. doi: 10.1136/thorax.55.3.210. No abstract available. PMID 10679540
- [Background] Dailloux M, Abalain ML, Laurain C, Lebrun L, Loos-Ayav C, Lozniewski A, Maugein J; French Mycobacteria Study Group. Respiratory infections associated with nontuberculous mycobacteria in non-HIV patients. Eur Respir J. 2006 Dec;28(6):1211-5. doi: 10.1183/09031936.00063806. PMID 17138678
- [Background] Jenkins PA, Campbell IA; Research Committee of The British Thoracic Society. Pulmonary disease caused by Mycobacterium xenopi in HIV-negative patients: five year follow-up of patients receiving standardised treatment. Respir Med. 2003 Apr;97(4):439-44. doi: 10.1053/rmed.2002.1444. PMID 12693807
- [Background] Baugnee PE, Pouthier F, Delaunois L. [Pulmonary mycobacteriosis due to Mycobacterium xenopi" in-vitro sensitivity to classical antitubercular agents and clinical development]. Acta Clin Belg. 1996;51(1):19-27. French. PMID 8669159
- [Background] Martin-Casabona N, Bahrmand AR, Bennedsen J, Thomsen VO, Curcio M, Fauville-Dufaux M, Feldman K, Havelkova M, Katila ML, Koksalan K, Pereira MF, Rodrigues F, Pfyffer GE, Portaels F, Urgell JR, Rusch-Gerdes S, Tortoli E, Vincent V, Watt B; Spanish Group for Non-Tuberculosis Mycobacteria. Non-tuberculous mycobacteria: patterns of isolation. A multi-country retrospective survey. Int J Tuberc Lung Dis. 2004 Oct;8(10):1186-93. PMID 15527150
- [Background] Yates MD, Pozniak A, Uttley AH, Clarke R, Grange JM. Isolation of environmental mycobacteria from clinical specimens in south-east England: 1973-1993. Int J Tuberc Lung Dis. 1997 Feb;1(1):75-80. PMID 9441063
- [Background] Andrejak C, Lescure FX, Douadi Y, Laurans G, Smail A, Duhaut P, Jounieaux V, Schmit JL. Non-tuberculous mycobacteria pulmonary infection: management and follow-up of 31 infected patients. J Infect. 2007 Jul;55(1):34-40. doi: 10.1016/j.jinf.2007.01.008. Epub 2007 Mar 13. PMID 17360040
- [Background] Andrejak C, Lescure FX, Pukenyte E, Douadi Y, Yazdanpanah Y, Laurans G, Schmit JL, Jounieaux V; Xenopi Group. Mycobacterium xenopi pulmonary infections: a multicentric retrospective study of 136 cases in north-east France. Thorax. 2009 Apr;64(4):291-6. doi: 10.1136/thx.2008.096842. Epub 2008 Dec 3. PMID 19052044
- [Background] Costrini AM, Mahler DA, Gross WM, Hawkins JE, Yesner R, D'Esopo ND. Clinical and roentgenographic features of nosocomial pulmonary disease due to Mycobacterium xenopi. Am Rev Respir Dis. 1981 Jan;123(1):104-9. doi: 10.1164/arrd.1981.123.1.104. PMID 7458072
- [Background] Andrejak C, Thomsen VO, Johansen IS, Riis A, Benfield TL, Duhaut P, Sorensen HT, Lescure FX, Thomsen RW. Nontuberculous pulmonary mycobacteriosis in Denmark: incidence and prognostic factors. Am J Respir Crit Care Med. 2010 Mar 1;181(5):514-21. doi: 10.1164/rccm.200905-0778OC. Epub 2009 Dec 10. PMID 20007929
- [Background] Dautzenberg B, Papillon F, Lepitre M, Truffot-Pernod C, Chauvin JP. Mycobacterium xenopi infections treated with clarithromycine-containing regimens. Annual meeting, 33rd Interscience Conference on Antimicrobial Agents and Chemotherapy.
- [Background] Alfandari S. Recommandations du C-CLIN Paris Nord pour le diagnostic et le traitement des infections ostéo-articulaires à Mycobacterium xenopi. Med Mal Infect 28 :231-234, 1998.
- [Background] Klemens SP, Cynamon MH. Activities of azithromycin and clarithromycin against nontuberculous mycobacteria in beige mice. Antimicrob Agents Chemother. 1994 Jul;38(7):1455-9. doi: 10.1128/AAC.38.7.1455. PMID 7979271
- [Background] Lounis N, Truffot-Pernot C, Bentoucha A, Robert J, Ji B, Grosset J. Efficacies of clarithromycin regimens against Mycobacterium xenopi in mice. Antimicrob Agents Chemother. 2001 Nov;45(11):3229-30. doi: 10.1128/AAC.45.11.3229-3230.2001. PMID 11600387
- [Background] Jenkins PA, Campbell IA, Banks J, Gelder CM, Prescott RJ, Smith AP. Clarithromycin vs ciprofloxacin as adjuncts to rifampicin and ethambutol in treating opportunist mycobacterial lung diseases and an assessment of Mycobacterium vaccae immunotherapy. Thorax. 2008 Jul;63(7):627-34. doi: 10.1136/thx.2007.087999. Epub 2008 Feb 4. PMID 18250184
- [Background] Varadi RG, Marras TK. Pulmonary Mycobacterium xenopi infection in non-HIV-infected patients: a systematic review. Int J Tuberc Lung Dis. 2009 Oct;13(10):1210-8. PMID 19793424
- [Background] Wallace RJ Jr, Brown BA, Griffith DE, Girard WM, Murphy DT. Clarithromycin regimens for pulmonary Mycobacterium avium complex. The first 50 patients. Am J Respir Crit Care Med. 1996 Jun;153(6 Pt 1):1766-72. doi: 10.1164/ajrccm.153.6.8665032.
- [Background] Dautzenberg B, Piperno D, Diot P, Truffot-Pernot C, Chauvin JP. Clarithromycin in the treatment of Mycobacterium avium lung infections in patients without AIDS. Clarithromycin Study Group of France. Chest. 1995 Apr;107(4):1035-40. doi: 10.1378/chest.107.4.1035. PMID 7705112
- [Background] Griffith DE, Brown BA, Cegielski P, Murphy DT, Wallace RJ Jr. Early results (at 6 months) with intermittent clarithromycin-including regimens for lung disease due to Mycobacterium avium complex. Clin Infect Dis. 2000 Feb;30(2):288-92. doi: 10.1086/313644. PMID 10671330
- [Background] Griffith DE, Brown BA, Girard WM, Murphy DT, Wallace RJ Jr. Azithromycin activity against Mycobacterium avium complex lung disease in patients who were not infected with human immunodeficiency virus. Clin Infect Dis. 1996 Nov;23(5):983-9. doi: 10.1093/clinids/23.5.983. PMID 8922790
- [Background] Tanaka E, Kimoto T, Tsuyuguchi K, Watanabe I, Matsumoto H, Niimi A, Suzuki K, Murayama T, Amitani R, Kuze F. Effect of clarithromycin regimen for Mycobacterium avium complex pulmonary disease. Am J Respir Crit Care Med. 1999 Sep;160(3):866-72. doi: 10.1164/ajrccm.160.3.9811086. PMID 10471610
- [Background] Dauendorffer JN, Laurain C, Weber M, Dailloux M. In vitro sensitivity of Mycobacterium xenopi to five antibiotics. Pathol Biol (Paris). 2002 Dec;50(10):591-4. doi: 10.1016/s0369-8114(02)00360-7. PMID 12504367
- [Background] Berlin OG, Young LS, Floyd-Reising SA, Bruckner DA. Comparative in vitro activity of the new macrolide A-56268 against mycobacteria. Eur J Clin Microbiol. 1987 Aug;6(4):486-7. doi: 10.1007/BF02013117. No abstract available. PMID 2959472
- [Background] Fraschini F, Scaglione F, Pintucci G, Maccarinelli G, Dugnani S, Demartini G. The diffusion of clarithromycin and roxithromycin into nasal mucosa, tonsil and lung in humans. J Antimicrob Chemother. 1991 Feb;27 Suppl A:61-5. doi: 10.1093/jac/27.suppl_a.61. PMID 1827103
- [Background] Wallace RJ Jr, Brown BA, Griffith DE. Drug intolerance to high-dose clarithromycin among elderly patients. Diagn Microbiol Infect Dis. 1993 Mar-Apr;16(3):215-21. doi: 10.1016/0732-8893(93)90112-k. PMID 8477575
- [Background] Gillespie SH, Billington O. Activity of moxifloxacin against mycobacteria. J Antimicrob Chemother. 1999 Sep;44(3):393-5. doi: 10.1093/jac/44.3.393. PMID 10511409
- [Background] Alcaide F, Calatayud L, Santin M, Martin R. Comparative in vitro activities of linezolid, telithromycin, clarithromycin, levofloxacin, moxifloxacin, and four conventional antimycobacterial drugs against Mycobacterium kansasii. Antimicrob Agents Chemother. 2004 Dec;48(12):4562-5. doi: 10.1128/AAC.48.12.4562-4565.2004. PMID 15561826
- [Background] Rodriguez Diaz JC, Lopez M, Ruiz M, Royo G. In vitro activity of new fluoroquinolones and linezolid against non-tuberculous mycobacteria. Int J Antimicrob Agents. 2003 Jun;21(6):585-8. doi: 10.1016/s0924-8579(03)00048-7. PMID 12791475
- [Background] Gosling RD, Uiso LO, Sam NE, Bongard E, Kanduma EG, Nyindo M, Morris RW, Gillespie SH. The bactericidal activity of moxifloxacin in patients with pulmonary tuberculosis. Am J Respir Crit Care Med. 2003 Dec 1;168(11):1342-5. doi: 10.1164/rccm.200305-682OC. Epub 2003 Aug 13. PMID 12917230
- [Background] Bermudez LE, Kolonoski P, Petrofsky M, Wu M, Inderlied CB, Young LS. Mefloquine, moxifloxacin, and ethambutol are a triple-drug alternative to macrolide-containing regimens for treatment of Mycobacterium avium disease. J Infect Dis. 2003 Jun 15;187(12):1977-80. doi: 10.1086/375352. Epub 2003 Jun 4. PMID 12792877
- [Background] Bermudez LE, Inderlied CB, Kolonoski P, Petrofsky M, Aralar P, Wu M, Young LS. Activity of moxifloxacin by itself and in combination with ethambutol, rifabutin, and azithromycin in vitro and in vivo against Mycobacterium avium. Antimicrob Agents Chemother. 2001 Jan;45(1):217-22. doi: 10.1128/AAC.45.1.217-222.2001. PMID 11120969
- [Background] Veziris N, Truffot-Pernot C, Aubry A, Jarlier V, Lounis N. Fluoroquinolone-containing third-line regimen against Mycobacterium tuberculosis in vivo. Antimicrob Agents Chemother. 2003 Oct;47(10):3117-22. doi: 10.1128/AAC.47.10.3117-3122.2003. PMID 14506018
- [Background] Valerio G, Bracciale P, Manisco V, Quitadamo M, Legari G, Bellanova S. Long-term tolerance and effectiveness of moxifloxacin therapy for tuberculosis: preliminary results. J Chemother. 2003 Feb;15(1):66-70. doi: 10.1179/joc.2003.15.1.66. PMID 12678417
- [Background] Moadebi S, Harder CK, Fitzgerald MJ, Elwood KR, Marra F. Fluoroquinolones for the treatment of pulmonary tuberculosis. Drugs. 2007;67(14):2077-99. doi: 10.2165/00003495-200767140-00007. PMID 17883288
- [Background] Shandil RK, Jayaram R, Kaur P, Gaonkar S, Suresh BL, Mahesh BN, Jayashree R, Nandi V, Bharath S, Balasubramanian V. Moxifloxacin, ofloxacin, sparfloxacin, and ciprofloxacin against Mycobacterium tuberculosis: evaluation of in vitro and pharmacodynamic indices that best predict in vivo efficacy. Antimicrob Agents Chemother. 2007 Feb;51(2):576-82. doi: 10.1128/AAC.00414-06. Epub 2006 Dec 4. PMID 17145798
- [Background] Teeter JG, Bleecker ER. Relationship between airway obstruction and respiratory symptoms in adult asthmatics. Chest. 1998 Feb;113(2):272-7. doi: 10.1378/chest.113.2.272. PMID 9498938
- [Background] Begaud B, Evreux JC, Jouglard J, Lagier G. [Imputation of the unexpected or toxic effects of drugs. Actualization of the method used in France]. Therapie. 1985 Mar-Apr;40(2):111-8. No abstract available. French. PMID 4002188
- [Background] Rhodes VA, McDaniel RW. The Index of Nausea, Vomiting, and Retching: a new format of the lndex of Nausea and Vomiting. Oncol Nurs Forum. 1999 Jun;26(5):889-94. PMID 10382187